CLINICAL TRIAL: NCT05638308
Title: Evaluation of Diagnostic Performance and Prognostic Value of 18F-Fluoroazomycin Arabinoside (FAZA) Positron Emission Tomography/Magnetic Resonance Imaging (PET/MR) in Patients With Kidney Graft Fibrosis
Brief Title: FAZA PETMRI Kidney Graft Fibrosis Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-5695
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Kidney Graft Fibrosis

STUDY DESIGN:
Intervention Model Description: FAZA PET/MRI Scan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAZA PET/MRI scan (Other): FAZA PET/MRI scan before the standard of care biopsy for case group
  Interventions: Diagnostic Test: FAZA PET/MRI scan

INTERVENTIONS:
Diagnostic Test: FAZA PET/MRI scan — FAZA PET/MRI scan before the standard of care biopsy for case group

SUMMARY:
Fibrosis is the final common pathway of solid organ diseases and accounts for ~45% of deaths in the developed world. Fibrosis is characterized by excessive deposition of extracellular matrix that replaces normal organ parenchyma, leading to loss of function. Chronic kidney disease is invariably characterized by fibrosis and affects >3 million Canadians. Although fibrosis can affect all compartments in the kidney. Interstitial fibrosis/tubular atrophy (IFTA) is the most potent predictor of kidney disease progression, regardless of its underlying cause. In addition to affecting native kidneys, IFTA also occurs in kidney allografts in transplanted patients, resulting in progressive kidney allograft dysfunction and, finally allograft loss with significant implications for patients' care and also financial implications for the healthcare system. However, early, noninvasive markers of IFTA or ongoing hypoxia in the kidney grafts are lacking. This is particularly problematic, since diagnosis of IFTA is often made late in the course of disease, and once IFTA develops, it is generally considered irreversible. There is thus an unmet clinical need to identify early markers of IFTA that could guide the use of novel anti-fibrotic therapies.

In patients with clinically decreasing allograft function or protienuria, indication (or for cause) biopsies are the gold standard test used to identify the cause for the functional decrease. However, biopsies carry significant procedural risk (e.g. bleeding and death) and suffer from a sampling bias - not all areas of the kidneys are accessible for biopsy and there is currently no way to target the fibrotic / hypoxic areas. Urine protein measurements are obviously also not suitable to resolve this clinical dilemma. There would thus be great clinical interest in developing non-invasive tools that could provide more information compared to traditional tests for monitoring renal hypoxia and injury through imaging and urinary biomarkers.

Our aims would be to image patients with different states of allograft function impairment and ideally find an imaging-based way to monitor those patients after transplantation. This way, an early detection of evolving interstitial fibrosis/tubular atrophy (IFTA) might be possible in a non-invasive way.The goal of this trial is to validate FAZA-PET/MR as a biomarker of hypoxia by correlating its uptake in patients with kidney allograft fibrosis with mass spectrometry based quantitative assays for monitoring of fibrotic markers in the urine of those same patients.

There would thus be great clinical interest in developing non-invasive tools that could provide more information compared to traditional tests for monitoring renal hypoxia and injury through imaging and urinary biomarkers. Whereas currently only allograft biopsy can be performed to detect (rather late stage) interstitial fibrosis/ tubular atrophy.

The study subjects' clinical management will not be changed based on the PET-MR scan within the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Evidence of impaired kidney graft function based on elevated serum creatinine from baseline and/ or evidence of significant proteinuria and/or donor specific antibodies
3. A negative urine or serum pregnancy test within the three week interval immediately prior to imaging, in women of child-bearing age
4. Ability to provide written informed consent to participate in the study (for both patients groups - with and without impaired kidney graft function)
5. Two study groups:

   * Evidence of impaired kidney graft function based on elevated serum creatinine from baseline and/ or evidence of significant proteinuria and/or donor specific antibodies and scheduled for a kidney graft biopsy.
   * comparison (control) group with stable kidney graft function, matched for graft/recipient age, sex and comorbidities

Exclusion Criteria:

1. Contraindication for MR as per current institutional guidelines
2. Inability to lie supine for at least 30 minutes
3. Any patient who is pregnant or breastfeeding
4. Any patient unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-26 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
To image patients with different states of allograft function impairment and ideally find an imaging-based way to monitor those patients after transplantation | Before the planned routine biopsy procedure for case patients
  The FAZA uptake during the PET/MRI scan
To image patients with different states of allograft function impairment and ideally find an imaging-based way to monitor those patients after transplantation | Through study completion once patient with stable graft function and minimal or no fibrosis on time zero biopsy and age matched graft age is identified. Up to 60 months
  The FAZA uptake during the PET/MRI scan

SECONDARY OUTCOMES:
Performing urine assays whereby AngII activity proteins in urine to predict the survival/viability outcome of the kidney allograft | Before the planned routine biopsy procedure for case patients
  Evaluate AngII-regulated proteins in urine samples
Performing urine assays whereby AngII activity proteins in urine to predict the survival/viability outcome of the kidney allograft | Through study completion once patient with stable graft function and minimal or no fibrosis on time zero biopsy and age matched graft age is identified. Up to 60 months
  Evaluate AngII-regulated proteins in urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Veit-Haibach, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada